CLINICAL TRIAL: NCT05632484
Title: Genotype Expression and Phenotype of Endothelial Cells, Carrying an ACVRL1, ENG or SMAD4 Mutation, in Response to BMP9 for the Identification of New Therapeutic Targets in Hereditary Haemorrhagic Telangiectasia
Acronym: CAERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL20_0250; 2021-A01792-39 (Other: ID-RCB)
Record Dates: First submitted 2022-10-21; First posted 2022-11-30 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Hereditary Haemorrhagic Telangiectasia
Keywords: hereditary haemorrhagic telangiectasia; endothelial cell
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Cordocentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Newborns with a parent with HHT disease (Experimental): 16 newborns with one parent suffering HHT disease and carrying a mutation in the ACVRL1, ENG or SMAD4 gene will be included in this study.
  Interventions: Biological: Cord blood sampling; Biological: Cord sampling

INTERVENTIONS:
Biological: Cord blood sampling — Collection of 2 milliliters (mL) of cord blood on an Ethylenediaminetetraacetic acid (EDTA) tube, on the day of delivery and after cutting the umbilical cord, for genetic testing
Biological: Cord blood sampling — Collection of 50 to 100 mL of cord blood from the cord blood collection bag
Biological: Cord sampling — Collection of 20 centimeters (cm) of umbilical cord

SUMMARY:
Hereditary hemorrhagic telangiectasia (HHT) or Osler-Weber-Rendu syndrome patients are carriers of a heterozygous mutation of the activin receptor-like kinase 1 (ACVRL1), Endoglin (ENG) or Mothers against decapentaplegic homolog 4 (SMAD4) gene. HHT involves the Bone Morphogenetic Protein 9 (BMP9)/Activin receptor-Like Kinase 1 (ALK1)-endoglin signalling pathway. BMP9 is a growth factor that binds to ALK1 receptor and to endoglin its co-receptors and physiologically activates Smad signaling pathway. Endothelial cells in HHT patients display half expression of functional ALK1 receptors or endoglin co-receptors or of the transcription factor SMAD4, which should lead to effects on the functions of these cells.

The identification of differences in gene expression between endothelial cells from HHT patients and healthy donors will allow the identification of new functions or new target pathways for therapy. Circulating endothelial cells are rare in the bloodstream in adults, but are present in greater quantities in cord blood.

ELIGIBILITY:
Inclusion Criteria:

* Newborn whose parents :

  * are adults
  * are affiliated to a social security or similar
  * are not subject to any legal protection measures
* Newborn child with one parent who has monitored for HHT confirmed by molecular biology (carrier of a mutation of the SMAD4, ENG or ACVRL1 gene).
* Consent signed by the two representatives of parental authority

Exclusion Criteria:

* One of the two parents opposes donating the umbilical cord blood and the umbilical cord for research
* One of the two parents opposes genetic testing
* Patient for whom it was not possible to obtain umbilical cord blood after delivery for technical or medical reasons.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Number of Endothelial Colony Forming Cells (ECFC) from cord blood | up to 3 weeks after cells isolation
  The primary outcome is the obtention of at least one clone of 10 000 cells from the cord blood after 3 weeks from the time of isolation. Number of viable cells is measured by Trypan blue test.
Number of Human Umbilical Vein Endothelial Cells(HUVEC) from cord | up to one week
  For the cord, the primary outcome is the obtention of 500 000 cells after one week from the isolation. Number of viable cells is measured by Trypan blue test.

SECONDARY OUTCOMES:
cell freezing and thawing | Through study completion, an average of 5 years.
  After isolation and amplification, cells from cord or from clones from the cord blood are frozen in vials. The cells viability (50 to 70% of alive cells after thawing) is a criteria of successful experiment.
Gene expression quantification after RNA extraction from cells | Through study completion, an average of 5 years.
  The third outcome is reached when we obtain up to 5 µg of RNA after cell seeding and stimulation with growth factors. Gene expression is measured by real-time polymerase chain reaction (RT-qPCR) and Ribonucleic acid Sequencing (RNAseq).

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Femme-mère-Enfant, Bron
  - Hôpital Estaing, Clermont-Ferrand
  - Hôpital St Eloi, Montpellier

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al Tabosh T, Al Tarrass M, Tourvieilhe L, Guilhem A, Dupuis-Girod S, Bailly S. Hereditary hemorrhagic telangiectasia: from signaling insights to therapeutic advances. J Clin Invest. 2024 Feb 15;134(4):e176379. doi: 10.1172/JCI176379. PMID 38357927
- [Background] Al Tabosh T, Liu H, Koca D, Al Tarrass M, Tu L, Giraud S, Delagrange L, Beaudoin M, Riviere S, Grobost V, Rondeau-Lutz M, Dupuis O, Ricard N, Tillet E, Machillot P, Salomon A, Picart C, Battail C, Dupuis-Girod S, Guignabert C, Desroches-Castan A, Bailly S. Impact of heterozygous ALK1 mutations on the transcriptomic response to BMP9 and BMP10 in endothelial cells from hereditary hemorrhagic telangiectasia and pulmonary arterial hypertension donors. Angiogenesis. 2024 May;27(2):211-227. doi: 10.1007/s10456-023-09902-8. Epub 2024 Jan 31. PMID 38294582